CLINICAL TRIAL: NCT03458858
Title: Berry Components and Blood Sugar & Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS59
Record Dates: First submitted 2018-01-03; First posted 2018-03-08 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mixed Berry Diet (Other): Participants will receive between 400 to 800 grams of mixed berries daily, as a proportion of their daily caloric intake added to their base diet. The base diet will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Interventions: Other: Mixed Berry Diet
- Carbohydrate Control Jello (Other): Participants will receive between 400 to 800 grams of strawberry jello daily, as a proportion of their daily caloric intake added to their base diet. The jello will be matched to the mixed berries in both total carbohydrate level and gram quantity. The base diet will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Interventions: Other: Carbohydrate Control Jello
- Fiber Enriched Jello (Other): Participants will receive between 400 to 800 grams of fiber enriched strawberry jello daily, as a proportion of their daily caloric intake added to their base diet. The jello will be matched to the mixed berries in both total carbohydrate level and fiber content, and in the same gram quantity. The base diet will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Interventions: Other: Fiber Enriched Jello
- Low Fiber Mixed Berry Juice (Other): Participants will receive 1 liter per day of low fiber mixed berry juice added to their base diet. The juice will be squeezed from the mixed berries, then filtered. The sugar level of the juice will match that of the mixed berries. The base diet will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Interventions: Other: Low Fiber Mixed Berry Juice

INTERVENTIONS:
Other: Mixed Berry Diet — Mixed Berry Treatment
  Arms: Mixed Berry Diet
Other: Carbohydrate Control Jello — Carbohydrate Control
  Arms: Carbohydrate Control Jello
Other: Fiber Enriched Jello — Fiber Control
  Arms: Fiber Enriched Jello
Other: Low Fiber Mixed Berry Juice — Anthocyanin Control
  Arms: Low Fiber Mixed Berry Juice

SUMMARY:
The primary objective of this study is to determine which components of berries improve glucose metabolism and increase fat oxidation in humans.

DETAILED DESCRIPTION:
The aim of this study is to improve understanding of how diet can regulate glucose metabolism and fuel use. Previous human and animal studies have demonstrated that berries can improve gluco-regulation and increase fat oxidation. The aim of this study is to determine which component of berries is conveying this health benefit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoker
* able to understand consent

Exclusion Criteria:

* Body Mass Index less than 25 kg/m2
* pregnant, lactating, having given birth in the past year
* allergy to berries
* blood glucose greater than 125 mg/dL
* history of bariatric surgery or nutrient malabsorption disease
* diagnosis or treatment of cancer in past three years
* type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Glucose Metabolism Phase 1 | Day 8
  Subjects will undergo a meal-based glucose tolerance test; blood samples will be analyzed for glucose in mmol/L.
Glucose Metabolism Phase 2 | Day 29
  Subjects will undergo a meal-based glucose tolerance test; blood samples will be analyzed for glucose in mmol/L.
Glucose Metabolism Phase 3 | Day 50
  Subjects will undergo a meal-based glucose tolerance test; blood samples will be analyzed for glucose in mmol/L.
Glucose Metabolism Phase 4 | Day 71
  Subjects will undergo a meal-based glucose tolerance test; blood samples will be analyzed for glucose in mmol/L.

SECONDARY OUTCOMES:
Insulin sensitivity | Day 8, 29, 50, 71
  Subjects will undergo a meal-based glucose tolerance test; blood samples will be analyzed for insulin in units of microIU/mL.
Fat trafficking | Day 8, 29, 50, 71
  Subjects will undergo a meal-based glucose tolerance test; blood samples will be analyzed for non-esterified fatty acids in mmol/L.
Peripheral mononuclear blood cells energetics | Day 8, 29, 50, 71
  Blood cells called peripheral mononuclear blood cells will be isolated and analyzed for mitochondrial function/oxygen consumption in nmol/ml.
Metabolic Fuel Use | Day 7-8, 28-29, 49-50, 70-71
  Subjects will spend the night in an indirect calorimeter to measure their oxygen consumption and carbon dioxide evolution which will be used to calculate the dietary energy source being oxidized, expressed as respiratory quotient which is a unitless ratio of liters of O2 inhaled to liters of CO2 exhaled.

OTHER OUTCOMES:
Metabolomics in blood | Day 8, 29, 50, 71
  Blood metabolomics profiling will be conducted by gas chromatography and liquid chromatography / time-of-flight mass spectrometry. Selected intensity of biochemicals in blood with mass ranging from 50 to 800 molecular weight will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No